CLINICAL TRIAL: NCT00715520
Title: Neurobiological Principles Applied to the Rehabilitation of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Cathrin Buetefisch, Dr. Cathrin Buetefisch, Emory University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00046953; R01NS060830-01A1 (NIH); NPARR01 (Other: Other)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Stroke
Keywords: Transcranial Magnetic Stimulation; Rehabilitation; Stroke; Plasticity
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; carbidopa, levodopa drug combination; Methylphenidate; Amphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aim 1 (Experimental): Healthy adult female and male subjects will receive study drugs and TMS training to measure M1 excitability.
  Interventions: Drug: Carbidopa-Levodopa; Drug: Methylphenidate; Drug: Amphetamine Sulfate; Drug: Placebo; Other: Transcranial Magnetic Stimulation (TMS) Training
- Aim 2 (Experimental): Healthy adult female and male subjects will receive repetitive TMS (rTMS) at different times or frequencies with respect to the training movement or sham stimulation.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS); Other: Sham Transcranial Magnetic Stimulation (TMS)
- Aim 3 (Experimental): Female and male subjects who have experienced a cerebral ischemic infarction, will receive study drugs and TMS to measure M1 excitability.
  Interventions: Drug: Carbidopa-Levodopa; Drug: Methylphenidate; Drug: Amphetamine Sulfate; Drug: Placebo; Other: Sham Transcranial Magnetic Stimulation (TMS); Other: Transcranial Magnetic Stimulation (TMS) Training

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — Each TMS training session will begin with a baseline measurement lasting about 30 minutes in which brief magnetic pulses will be generated by the single-pulse and paired pulse TMS stimulator and the responses are recorded with surface EMG electrodes. Participants will be instructed to move their wrist for up to ½ hour. After these measures, rTMS will be applied to the scalp during training. Stimulation will occur at a low rate of different frequencies and different times with respect to the training movement depending on the experimental condition. In the last phase of the session post-training measurements will be done using single TMS pulses. TMS pulses and intensity with be given in random order.
  Arms: Aim 2
Drug: Carbidopa-Levodopa — Participants will receive one oral dose of carbidopa-levodopa 25mg one hour prior to measuring wrist extension movements.
  The order in which Carbidopa-Levodopa is given will be randomized per participant.
  Other Names: Sinemet
  Arms: Aim 1; Aim 3
Drug: Methylphenidate — Participants will receive one oral dose of methylphenidate 40mg 2 hours prior to measuring wrist extension movements.
  The order in which Methylphenidate is given will be randomized per participant.
  Arms: Aim 1; Aim 3
Drug: Amphetamine Sulfate — Participants will receive one oral dose of amphetamine sulfate 10mg 2 hours prior to measuring wrist extension movements.
  The order in which Amphetamine Sulfate is given will be randomized per participant.
  Arms: Aim 1; Aim 3
Drug: Placebo — Participants will receive one oral tablet of placebo 2 hours prior to measuring wrist extension movements.
  The order in which Placebo is given will be randomized per participant.
  Arms: Aim 1; Aim 3
Other: Sham Transcranial Magnetic Stimulation (TMS) — Sham TMS pulses will be randomly administered during TMS sessions.
  Arms: Aim 2; Aim 3
Other: Transcranial Magnetic Stimulation (TMS) Training — TMS surface electromyographic activity will be recorded with surface electrodes mounted on the skin overlaying a forearm muscle. Single pulses of TMS at increasing intensity will be delivered to measure motor cortex excitability. Peak acceleration and TMS evoked responses in the muscle will be measured prior to the training, after completion of the training and again one hour after completion of the training.
  Arms: Aim 1; Aim 3

SUMMARY:
The purpose of this study is to use (Transcranial Magnetic Stimulation) TMS or drugs to improve learning of movement skills and the adaptation processes in patients after stroke. Once investigators have determined the improving effect of TMS and the drugs on learning of movement skills, the study team may be able to provide information that improves rehabilitative treatment and helps to improve recovery after stroke.

DETAILED DESCRIPTION:
Previous studies have shown, that when patients learn a new motor movement, it may cause a change in the way the nerves act in the area of the brain that controls movement. This change is called use-dependent plasticity. The ability of that part of the brain, called the motor cortex (M1), to reorganize plays a major role in the recovery of motor deficits post-stroke; hence the importance for further development of rehabilitative strategies that utilize this potential for recovery. In this proposed study, investigators will further examine influences of use-dependent plasticity in the non-injured M1 of healthy subjects and injured M1 of stroke subjects using a combination of non-invasive cortical stimulation, medication, and exercise techniques. In Aim 1, investigators will test the effect of drugs that interact specifically with different neurotransmitter systems on use-dependent plasticity in intact M1 of healthy humans. In Aim 2, investigators will identify the parameters for non-invasive transcranial magnetic stimulation (TMS) of M1 that are most effective to enhance use-dependent plasticity in intact healthy human M1. In Aim 3, investigators will test the drugs and rTMS protocols that were demonstrated to be most effective to enhance use- dependent plasticity in the Specific Aim 1 and 2 and apply them to participants who have experienced a stroke. Results from this study will help to inform future research about the efficacy of plasticity enhancing methods in injured M1 of stroke patients.

ELIGIBILITY:
Aims 1 and 2

Inclusion Criteria:

* Normal neurological examination
* Ability to meet criteria of inclusion experiment
* Ability to give informed consent.

Exclusion Criteria:

* History or neurological or psychiatric disease
* Abnormal MRI of brain
* Abnormal neuropsychological testing
* Intake of CNS active drugs
* History of seizure disorder
* History of migraine headaches
* History of anaphylaxis or allergic reactions
* Contraindication to TMS

Aim 3:

Inclusion Criteria:

* Cerebral ischemic infarction more than 6 months prior to entering the study
* Single lesion as defined by MRI of the brain affecting the primary motor output system of the hand at a cortical (M1) level or subcortical level, or unilateral, and supratentorial in absence of history of a previous symptomatic stroke within 3 months of the current stroke
* Dense paresis of the hand for more than three days after cerebral infarction (MRC of < 4- of wrist- and finger extension/flexion movements)
* Good functional recovery of hand function as defined by MRC of 4 or 4+ of wrist- and finger extension/flexion movements
* Ability to perform wrist extension movements
* Ability to meet criteria of inclusion experiment
* Ability to give informed consent
* Ability of TMS to elicit a measurable MEP of > 100 μV and an increase in MEP amplitude with increasing stimulus intensity (up to 100% of MSO) of at least 20% over MEP amplitude at MT

Exclusion Criteria:

* History or neurological or psychiatric disease, including bipolar disorder
* Intake of CNS active drugs
* History of seizure disorder
* History of migraine headaches
* History of anaphylaxis or allergic reactions
* Contraindication to TMS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin M Buetefisch, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 2007 and August 2013.
Groups:
- Aim 1: Healthy adult female and male subjects received study drugs and TMS to measure M1 excitability.
- Aim 2: Healthy adult female and male subjects received TMS prior to measuring wrist extension movements.
- Aim 3: Female and male subjects who have experienced a cerebral ischemic infarction will receive study drugs and TMS to measure M1 excitability.
Period: Overall Study
Arm/Group | Aim 1 | Aim 2 | Aim 3
Started | 20 | 10 | 3
Completed | 10 | 9 | 1
Not Completed | 10 | 1 | 2
Not completed — Screen failure | 8 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants included in the baseline analysis received a study intervention and completed all study procedures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 1 | Aim 2 | Aim 3 | Total
Number analyzed (Participants) | 10 | 9 | 1 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 1 | 15
  >=65 years | 3 | 2 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 1 | 12
  Male | 5 | 3 | 0 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 1 | 20

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Mean Parameter Estimate for Maximal Motor Evoked Potential (MEPmax) Derived From Stimulus Response Curves (SRC)
Description: Motor evoked potential (MEP) amplitudes were measured prior to treatment (baseline), immediately after the treatment (post-training 1), 30 minutes after the treatment (post-training 2), and 60 minutes after the treatment (post-training 3).The MEP is elicited by transcranial magnetic stimulation (TMS) at increased intensity. Its amplitude is measured from peak to peak and expressed in millivolts (mV). Measured MEP amplitudes were plotted against the intensity to create a stimulus response curve (SRC). SRCs were modeled by a 3- parameter sigmoid function and MEPmax was extracted. Long-lasting increases in MEP amplitude indicate increases in motor cortex excitability and are associated with motor learning.
Time Frame: Baseline, Post-Training 1 (Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: Analysis was completed in Aim 1 participants per protocol for the placebo condition. One subject was not included in the analysis due to corrupt data.
Measure: Mean (Standard Error); unit: mV
Arm/Group | Aim 1
Number analyzed (Participants) | 9
mV
  Baseline Placebo - MEPmax | 1.01 (.13)
  Post-Training 1 Placebo - MEPmax | 1.63 (.33)
  Post-Training 2 Placebo - MEPmax | 1.29 (.05)
  Baseline - Amphetamine Sulfate - MEPmax | .73 (.10)
  Post-Training 1 Ampletamine Sulfate - MEPmax | 1.22 (.26)
  Post-Training 2 Amphetamine Sulfate - MEPmax | 1.08 (.04)
  Baseline Methylphenidate - MEPmax | 1.04 (.13)
  Post-Training 1 Methylphenidate - MEPmax | 1.10 (.12)
  Post-Training 2 Methylphenidate - MEPmax | 1.22 (.06)
  Baseline Carbidopa-Levodopa - MEPmax | 1.81 (.62)
  Post-Training 1 Carbidopa-Levodopa - MEPmax | 1.41 (.26)
  Post-Training 2 Carbidopa-Levodopa - MEPmax | 1.53 (.13)

2. Primary Outcome: Aim 1: Mean Peak Acceleration of Wrist Extension Movements
Description: Mean peak acceleration was measured across study drug conditions prior to treatment (baseline), immediately after the treatment (post-training 1), 30 minutes after the treatment (post-training 2) and 60 minutes after the treatment (post-training 3). Increases in the mean peak acceleration of the trained wrist extension movements indicate motor learning. Acceleration was measured in g; a symbol for the average acceleration produced by gravity at the Earth's surface.
Time Frame: Baseline, Post-Training 1 (Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: Analysis was completed in Aim 1 participants per protocol. One subject was not included in the analysis due to corrupt data.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Aim 1
Number analyzed (Participants) | 9
g
  Baseline - Placebo | 1.32 (.35)
  Post-Training 1 - Placebo | 1.33 (.21)
  Post-Training 2 - Placebo | 1.24 (.30)
  Baseline - Amphetamine Sulfate | 1.24 (.33)
  Post-Training 1 - Amphetamine Sulfate | 1.28 (.31)
  Post-Training 2 - Amphetamine Sulfate | 1.29 (.39)
  Baseline - Methylphenidate | 1.35 (.30)
  Post-Training 1 - Methylphenidate | 1.27 (.16)
  Post-Training 2 - Methylphenidate | 1.22 (.25)
  Baseline - Carbidopa-Levodopa | 1.22 (.39)
  Post-Training 1 - Carbidopa-Levodopa | 1.23 (.27)
  Post-Training 2 - Carbidopa-Levodopa | 1.37 (.38)

3. Secondary Outcome: Aim 2: Mean Sum of Normalized Motor Evoked Potentials (MEPs) With Respect to Pulse
Description: Mean sum of normalized MEP for repeated TMS (rTMS) conditions with respect to the pulse (-100, +300, placebo, zero) prior to treatment (baseline), immediately after the treatment (post-training 1), 30 minutes after the treatment (post-training 2) and 60 minutes after the treatment (post-training 3). Its amplitude is measured from peak to peak and expressed in mV. Long- lasting increases in MEP amplitude indicate increases in motor cortex excitability and are associated with motor learning.
Time Frame: Baseline, Post-Training 1(Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: Analysis was completed in Aim 2 participants per protocol.
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Aim 2
Number analyzed (Participants) | 9
millivolts
  Baseline - Pulse (zero) | .39 (.36)
  Post-Training 1 - Pulse (zero) | .66 (.74)
  Post-Training 2 - Pulse (zero) | .63 (.63)
  Post-Training 3 - Pulse (zero) | .69 (.76)
  Baseline - Pulse (placebo) | .40 (.38)
  Post-Training 1 - Pulse (placebo) | .54 (.57)
  Post-Training 2 - Pulse (placebo) | .51 (.59)
  Post-Training 3 - Pulse (placebo) | .52 (.59)
  Baseline - Pulse (-100) | .39 (.37)
  Post-Training 1 - Pulse (-100) | .56 (.54)
  Post-Training 2 - Pulse (-100) | .60 (.67)
  Post-Training 3 - Pulse (-100) | .61 (.63)
  Baseline - Pulse (+300) | .38 (.38)
  Post-Training 1 - Pulse (+300) | .54 (.51)
  Post-Training 2 - Pulse (+300) | .48 (.45)
  Post-Training 3 - Pulse (+300) | .51 (.50)

4. Secondary Outcome: Aim 2: Mean Peak Acceleration of Wrist Extension Movements With Respect to Pulse
Description: Mean peak acceleration of wrist movements for repeated TMS (rTMS) conditions with respect of the TMS pulse (-100, +300, placebo, zero) prior to treatment (baseline), immediately after the treatment (post-training 1), 30 minutes after the treatment (post-training 2) and 60 minutes after the treatment (post-training 3). Increases in the mean peak acceleration of the trained wrist extension movements indicate motor learning. Acceleration was measured in g; a symbol for the average acceleration produced by gravity at the Earth's surface.
Time Frame: Baseline, Post-Training 1(Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: Analysis was completed in Aim 2 participants per protocol.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Aim 2
Number analyzed (Participants) | 9
g
  Baseline - Pulse (zero) | 1.33 (.31)
  Post-Training 1 - Pulse (zero) | 1.43 (.30)
  Post-Training 2 - Pulse (zero) | 1.51 (.34)
  Post-Training 3 - Pulse (zero) | 1.53 (.37)
  Baseline - Pulse (placebo) | 1.44 (.25)
  Post-Training 1 - Pulse (placebo) | 1.36 (.24)
  Post-Training 2 - Pulse (placebo) | 1.35 (.24)
  Post-Training 3 - Pulse (placebo) | 1.33 (.30)
  Baseline - Pulse (-100) | 1.51 (.34)
  Post-Training 1 - Pulse (-100) | 1.5 (.30)
  Post-Training 2 - Pulse (-100) | 1.46 (.34)
  Post-Training 3 - Pulse (-100) | 1.47 (.27)
  Baseline - Pulse (+300) | 1.40 (.34)
  Post-Training 1 - Pulse (+300) | 1.32 (.35)
  Post-Training 2 - Pulse (+300) | 1.38 (.40)
  Post-Training 3 - Pulse (+300) | 1.40 (.43)

5. Secondary Outcome: Aim 2: Mean Sum of Normalized Motor Evoked Potentials (MEPs) for rTMS Treatment With Respect to Frequency
Description: Mean sum of normalized MEP for the different frequencies of rTMS treatment (placebo at 0.1 Hz, 0.1 Hz, 0.25 Hz, 0.5 Hz) prior to treatment (baseline), immediately after the treatment (post-training 1), 30 minutes after the treatment (post-training 2) and 60 minutes after the treatment (post-training 3). Increases in the mean peak acceleration of the trained wrist extension movements indicate motor learning.
Time Frame: Baseline, Post-Training 1(Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: Analysis was completed in Aim 2 participants per protocol.
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Aim 2
Number analyzed (Participants) | 9
millivolts
  Baseline - Placebo | .67 (.79)
  Post-Training 1 - Placebo | .93 (1.00)
  Post-Training 2 - Placebo | .94 (1.09)
  Post-Training 3 - Placebo | 1.02 (1.19)
  Baseline - .1 Hz | .71 (.83)
  Post-Training 1 - .1 Hz | 1.06 (1.15)
  Post-Training 2 - .1 Hz | 1.06 (1.23)
  Post-Training 3 - .1 Hz | 1.14 (1.24)
  Baseline - .25 Hz | .67 (.84)
  Post-Training 1 - .25 Hz | .90 (1.03)
  Post-Training 2 - .25 Hz | .90 (1.08)
  Post-Training 3 - .25 Hz | .98 (1.15)
  Baseline - .5 Hz | .64 (.74)
  Post-Training 1 - .5 Hz | .92 (1.11)
  Post-Training 2 - .5 Hz | .90 (.99)
  Post-Training 3 - .5 Hz | .84 (1.00)

6. Secondary Outcome: Aim 2: Mean Peak Acceleration for rTMS Treatment With Respect to Frequency
Description: Mean peak acceleration for the different frequencies of rTMS treatment (placebo, 0.1 Hz, 0.25 Hz, 0.5 Hz) prior to treatment (baseline), immediately after the treatment (post-training 1), 30 minutes after the treatment (post-training 2) and 60 minutes after the treatment (post-training 3). Increases in the mean peak acceleration of the trained wrist extension movements indicate motor learning. Acceleration was measured in g; a symbol for the average acceleration produced by gravity at the Earth's surface.
Time Frame: Baseline, Post-Training 1(Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: Analysis was completed in Aim 2 participants per protocol.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Aim 2
Number analyzed (Participants) | 9
g
  Baseline - Placebo | 1.44 (.25)
  Post-Training 1 - Placebo | 1.36 (.24)
  Post-Training 2 - Placebo | 1.35 (.24)
  Post-Training 3 - Placebo | 1.33 (.30)
  Baseline - .1 Hz | 1.33 (.31)
  Post-Training 1 - .1 Hz | 1.43 (.30)
  Post-Training 2 - .1 Hz | 1.50 (.34)
  Post-Training 3 - .1 Hz | 1.53 (.37)
  Baseline - .25 Hz | 1.38 (.26)
  Post-Training 1 - .25 Hz | 1.35 (.44)
  Post-Training 2 - .25 Hz | 1.40 (.37)
  Post-Training 3 - .25 Hz | 1.34 (.47)
  Baseline - .5 Hz | 1.32 (.23)
  Post-Training 1 - .5 Hz | 1.29 (.30)
  Post-Training 2 - .5 Hz | 1.25 (.29)
  Post-Training 3 - .5 Hz | 1.29 (.31)

7. Secondary Outcome: Aim 3: Mean Parameter Estimate for Maximal Motor Evoked Potential (MEPmax) Derived From Stimulus Response Curves (SRC)
Description: as for outcome 1
Time Frame: Baseline, Post-Training 1(Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: No sufficient data collected.
Arm/Group | Aim 3
Number analyzed (Participants) | 0

8. Secondary Outcome: Aim 3: Mean Peak Acceleration of Wrist Extension Movements
Description: as for outcome 2
Time Frame: Baseline, Post-Training 1(Immediately), Post-Training 2 (30 Minutes), Post-Training 3 (60 Minutes)
Population: No sufficient data collected.
Arm/Group | Aim 3
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (6 years, 6 months).
Arm/Group | Aim 1 | Aim 2 | Aim 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/1
Other Adverse Events (participants affected / at risk) | 5/10 | 0/9 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aim 1 (N=10) | Aim 2 (N=9) | Aim 3 (N=1)
Vertio (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Increased Blood Pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parathesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial Edema (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Target enrollment for aim 3 was not me due to difficulty identifying participants that met the inclusion criteria. Therefore the study team did not have a sufficient sample size to complete any data analysis for this aim.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes